CLINICAL TRIAL: NCT07268703
Title: Effect of Expiratory Muscle Strength Training in Patients With Parkinson's Disease and Forward Trunk Flexion: A Pilot Study
Brief Title: Expiratory Muscle Training in Parkinson's Disease With Forward Trunk Flexion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Kateřina Dvořáková, Physiotherapist, General University Hospital, Prague
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45-25 S-IV
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Expiratory Muscle Strength Training; Forward Trunk Flexion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD with Forward Trunk Flexion (Experimental): Participants in this arm have Parkinson's disease and forward trunk flexion, defined as thoracic flexion ≥25° or lumbar flexion ≥15° while standing and walking, which completely disappears when lying down.
  They will follow the study schedule including all assessments and the 4-week EMST program. Outcomes will include voluntary peak cough flow, respiratory muscle strength, swallowing function (FEES), drooling, and posture assessment using standardized photographs.
  Interventions: Device: Expiratory muscle strength training
- PD without Forward Trunk Flexion (Active Comparator): Participants in this arm have Parkinson's disease without forward trunk flexion (no postural abnormalities).
  They will follow the same study schedule including all assessments and the 4-week EMST program as the experimental group.
  Interventions: Device: Expiratory muscle strength training

INTERVENTIONS:
Device: Expiratory muscle strength training — Participants will perform a 4-week Expiratory Muscle Strength Training (EMST) program using the EMST150™ device. EMST therapy sessions will be completed at home on 5 days per week, at the participant's convenience, performing five sets of five forceful exhalations through the device. The resistance of the device will be set to 75% of the patient's individual maximum expiratory pressure (MEP). The daily training will take approximately 15 minutes. Device resistance will be recalibrated at visits in weeks 0, 2, and 4 to ensure correct training and settings.

SUMMARY:
Postural abnormalities (PA) negatively affecting the axial system are part of the symptoms of Parkinson's disease (PD). They occur in more than 20% of patients with PD especially in more advanced stages of the disease, contribute significantly to patient disability, affect respiratory functions, and reduce quality of life. Eighty-five percent of patients with forward trunk flexion (FTF) reported difficulties with swallowing (dysphagia), shortness of breath, and drooling. Previous studies in patients with PD also identified cough disorders (dystussia). Since cough and properly functioning swallowing are key mechanisms for airway protection, impairments in these functions lead to a higher risk of aspiration. The seriousness of this problem is clearly confirmed by the fact that aspiration pneumonia is the leading cause of death in patients with PD.

Among non-pharmacological interventions for airway protection, expiratory muscle strength training (EMST) has been shown to be beneficial in patients with PD. Recent randomized controlled studies demonstrated a significant effect of EMST on dysphagia, dystussia, drooling, and dysarthria in patients with PD.

However, the literature lacks data on the effect of EMST on dystussia in patients with PD and FTF, who, according to previous research, are also affected by restrictive ventilatory impairment, which negatively affects respiratory capacity and, in particular, cough strength.

The aim of this study is to evaluate the effect of EMST on cough, swallowing, respiratory muscle strength, and drooling in patients with PD and forward trunk flexion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson' s disease
* Age ≥ 18 years
* MoCA score (Montreal Cognitive Assessment) ≥ 19
* Score II-IV during the "ON" phase under regular antiparkinsonian medication according to the Modified Hoehn and Yahr Scale
* Pathological forward trunk flexion defined as thoracic (≥ 25°) or lumbar flexion (> 15°) during standing and walking, which completely disappears in the supine position (for the experimental group only)

Exclusion Criteria:

* Change in antiparkinsonian medication within the last 3 months prior to study enrollment
* Other neurological, orthopedic, cardiovascular, or respiratory comorbidities
* Inability to cooperate due to neuropsychological dysfunction
* Current smoking history
* Inadequate lip seal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Voluntary peak cough flow | Week -1, week 0, week 4, week 8
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

SECONDARY OUTCOMES:
Assessment of Swallowing | Week -1, week 4, week 8
  Swallowing will be assessed using a flexible endoscopic evaluation of swallowing (FEES). This is a standardized examination of the swallowing process, which involves transnasal insertion of a flexible endoscope into the pharynx, followed by evaluation of food passage. The assessment will be performed according to established protocols for patients with Parkinson's disease. All FEES examinations will be video-recorded, anonymized, and subsequently independently evaluated by blinded raters in a randomized order.
Assessment of Drooling | Week -1, week 4, week 8
  Drooling will be assessed using a questionnaire consisting of seven items evaluating the presence and severity of uncontrolled saliva leakage from the mouth in various aspects of daily life in patients with Parkinson's disease.
Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) | Week -1, week 0, week 4, week 8
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Forced vital capacity (FVC) | Week -1, week 0, week 4, week 8
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Forced expiratory volume (FEV1) | Week -1, week 0, week 4, week 8
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Peak expiratory flow (PEF) | Week -1, week 0, week 4, week 8
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Tinazzi M, Geroin C, Bhidayasiri R, Bloem BR, Capato T, Djaldetti R, Doherty K, Fasano A, Tibar H, Lopiano L, Margraf NG, Merello M, Moreau C, Ugawa Y, Artusi CA; International Parkinson and Movement Disorders Society Task Force on Postural Abnormalities. Task Force Consensus on Nosology and Cut-Off Values for Axial Postural Abnormalities in Parkinsonism. Mov Disord Clin Pract. 2022 May 9;9(5):594-603. doi: 10.1002/mdc3.13460. eCollection 2022 Jul. PMID 35844289
- [Background] Forsyth AL, Joshi RY, Canning CG, Allen NE, Paul SS. Flexed Posture in Parkinson Disease: Associations With Nonmotor Impairments and Activity Limitations. Phys Ther. 2019 Jul 1;99(7):893-903. doi: 10.1093/ptj/pzz033. PMID 30830153
- [Background] Troche MS, Rosenbek JC, Okun MS, Sapienza CM. Detraining outcomes with expiratory muscle strength training in Parkinson disease. J Rehabil Res Dev. 2014;51(2):305-10. doi: 10.1682/JRRD.2013.05.0101. PMID 24933728
- [Background] Cocks N, Rafols J, Embley E, Hill K. Expiratory Muscle Strength Training for Drooling in Adults with Parkinson's Disease. Dysphagia. 2022 Dec;37(6):1525-1531. doi: 10.1007/s00455-022-10408-6. Epub 2022 Feb 16. PMID 35171321
- [Background] Claus I, Muhle P, Czechowski J, Ahring S, Labeit B, Suntrup-Krueger S, Wiendl H, Dziewas R, Warnecke T. Expiratory Muscle Strength Training for Therapy of Pharyngeal Dysphagia in Parkinson's Disease. Mov Disord. 2021 Aug;36(8):1815-1824. doi: 10.1002/mds.28552. Epub 2021 Mar 2. PMID 33650729
- [Background] Troche MS, Curtis JA, Sevitz JS, Dakin AE, Perry SE, Borders JC, Grande AA, Mou Y, Vanegas-Arroyave N, Hegland KW. Rehabilitating Cough Dysfunction in Parkinson's Disease: A Randomized Controlled Trial. Mov Disord. 2023 Feb;38(2):201-211. doi: 10.1002/mds.29268. Epub 2022 Nov 7. PMID 36345090
- [Background] Margraf NG, Granert O, Hampel J, Wrede A, Schulz-Schaeffer WJ, Deuschl G. Clinical Definition of Camptocormia in Parkinson's Disease. Mov Disord Clin Pract. 2016 Oct 11;4(3):349-357. doi: 10.1002/mdc3.12437. eCollection 2017 May-Jun. PMID 30363363
- [Background] Tinazzi M, Gandolfi M, Ceravolo R, Capecci M, Andrenelli E, Ceravolo MG, Bonanni L, Onofrj M, Vitale M, Catalan M, Polverino P, Bertolotti C, Mazzucchi S, Giannoni S, Smania N, Tamburin S, Vacca L, Stocchi F, Radicati FG, Artusi CA, Zibetti M, Lopiano L, Fasano A, Geroin C. Postural Abnormalities in Parkinson's Disease: An Epidemiological and Clinical Multicenter Study. Mov Disord Clin Pract. 2019 Jun 29;6(7):576-585. doi: 10.1002/mdc3.12810. eCollection 2019 Sep. PMID 31538092